CLINICAL TRIAL: NCT04250727
Title: Switching to a Non-tobacco-based Oral Nicotine Product Among Adult Cigarette Smokers: Exploring the Roles of Product Characteristics and User History
Brief Title: Switching to Potential Reduced Exposure Products in Adult Smokers
Acronym: ZYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2000023826
Record Dates: First submitted 2020-01-17; First posted 2020-01-31 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Tobacco Use Disorder; Oral Nicotine Pouch Use; Smoking Behaviors; Harm Reduction; Toxic Effect of Tobacco and Nicotine; Carcinogenesis
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Harm Reduction; Carcinogenesis

STUDY DESIGN:
Intervention Model Description: 30 current non-treatment seeking adult smokers will be randomized to either the 3mg or 6mg nicotine concentration ZYN condition.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3mg Nicotine Concentration (Experimental): 15 participants will be randomly assigned to receive ZYN Pouches with 3mg nicotine concentration.
  Interventions: Device: ZYN
- 6mg Nicotine Concentration (Experimental): 15 participants will be randomly assigned to receive ZYN Pouches with 6mg nicotine concentration.
  Interventions: Device: ZYN

INTERVENTIONS:
Device: ZYN — 30 current non-treatment seeking adult smokers will be switched from smoking cigarettes to ZYN oral nicotine pouches containing either 3mg or 6mg concentration nicotine salts.

SUMMARY:
This study aims to assess the feasibility, acceptability, and the potential harm reduction of switching to potentially lower risk, oral nicotine pouches in adult smokers. Part One of this study aims to assess the interest of current smokers in switching to an e-cigarette device (i.e. JUUL) compared to alternative non-combustible tobacco products (i.e. smokeless tobacco/snus) and/or medicinal nicotine via survey. Part Two will consist of a pilot study of 30 non-treatment seeking adult smokers to investigate within-person changes in smoking behavior as a result of switching to different concentrations of oral nicotine pouch products (i.e. ZYN, 3mg and 6mg nicotine concentration). Additionally, by measuring bio-markers of tobacco exposure from baseline, this will allow the study to assess the potential for harm reduction in switching from cigarettes to oral nicotine pouches.

ELIGIBILITY:
Inclusion Criteria:

1. 21-77 years old(in line with NIH guidelines for 18+ being the age of consent in adults) (2008 PHS Guideline Update Panel)
2. English literate
3. Smoke at least 1 cigarette per day
4. Expired breath carbon monoxide level ≥ 6ppm at baseline
5. Not currently actively pursuing smoking cessation services or planning to use evidence-based cessation tools to quit in the next month
6. Not interested in the use of existing FDA-approved tobacco pharmacotherapies (i.e., NRT, wellbutrin, varenicline).

Exclusion Criteria:

1. Currently using any stop smoking treatments (2008 PHS Guideline Update Panel)
2. History of serious psychiatric condition (i.e., bipolar disorder, schizophrenia)
3. Current uncontrolled medical condition
4. Cardiac conditions that required a hospitalization or intensive treatment on an outpatient basis in the past year including: myocardial infarction, coronary artery disease, unstable angina, congestive heart failure, or tachyarrhythmias (including rapid atrial fibrillation, ventricular tachycardia, or ventricular fibrillation)
5. Female participants of child-bearing age will be excluded if they are currently pregnant or breastfeeding or report an unwillingness to use effective birth control (i.e., abstinence, IUD, implant, sterilization, pill, patch, ring, or barrier method such as condoms) for the duration of the study
6. Severe lung disease that requires supplemental oxygen
7. Uncontrolled asthma (<20 on the Asthma Control Test (ACT) or requiring steroids more than 1x per year)
8. Unstable COPD: defined as GOLD category C or D (more than 2 exacerbations or 1 exacerbation leading to hospitalization in the past year)
9. Planning to quit smoking with a set goal or time for quit attempt
10. Known hypersensitivity to propylene glycol
11. Patients with an FEV1 < 40%

Ages: 21 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berg CJ, Haardoerfer R, Escoffery C, Zheng P, Kegler M. Cigarette users' interest in using or switching to electronic nicotine delivery systems for smokeless tobacco for harm reduction, cessation, or novelty: a cross-sectional survey of US adults. Nicotine Tob Res. 2015 Feb;17(2):245-55. doi: 10.1093/ntr/ntu103. Epub 2014 Jun 20. PMID 24951496
- [Background] Brawley OW, Glynn TJ, Khuri FR, Wender RC, Seffrin JR. The first Surgeon General's report on smoking and health: the 50th anniversary. CA Cancer J Clin. 2014 Jan-Feb;64(1):5-8. doi: 10.3322/caac.21210. Epub 2013 Nov 18. No abstract available. PMID 24249254
- [Background] Brenner DR, Scherer D, Muir K, Schildkraut J, Boffetta P, Spitz MR, Le Marchand L, Chan AT, Goode EL, Ulrich CM, Hung RJ. A review of the application of inflammatory biomarkers in epidemiologic cancer research. Cancer Epidemiol Biomarkers Prev. 2014 Sep;23(9):1729-51. doi: 10.1158/1055-9965.EPI-14-0064. Epub 2014 Jun 24. PMID 24962838
- [Background] Cappelleri JC, Bushmakin AG, Baker CL, Merikle E, Olufade AO, Gilbert DG. Confirmatory factor analyses and reliability of the modified cigarette evaluation questionnaire. Addict Behav. 2007 May;32(5):912-23. doi: 10.1016/j.addbeh.2006.06.028. Epub 2006 Jul 27. PMID 16875787
- [Background] Cella D, Lai JS, Jensen SE, Christodoulou C, Junghaenel DU, Reeve BB, Stone AA. PROMIS Fatigue Item Bank had Clinical Validity across Diverse Chronic Conditions. J Clin Epidemiol. 2016 May;73:128-34. doi: 10.1016/j.jclinepi.2015.08.037. Epub 2016 Mar 3. PMID 26939927
- [Background] Chang CM, Edwards SH, Arab A, Del Valle-Pinero AY, Yang L, Hatsukami DK. Biomarkers of Tobacco Exposure: Summary of an FDA-Sponsored Public Workshop. Cancer Epidemiol Biomarkers Prev. 2017 Mar;26(3):291-302. doi: 10.1158/1055-9965.EPI-16-0675. Epub 2016 Nov 9. PMID 28151705
- [Background] Jamal A, Phillips E, Gentzke AS, Homa DM, Babb SD, King BA, Neff LJ. Current Cigarette Smoking Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Jan 19;67(2):53-59. doi: 10.15585/mmwr.mm6702a1. PMID 29346338
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Background] Delnevo CD, Giovenco DP, Steinberg MB, Villanti AC, Pearson JL, Niaura RS, Abrams DB. Patterns of Electronic Cigarette Use Among Adults in the United States. Nicotine Tob Res. 2016 May;18(5):715-9. doi: 10.1093/ntr/ntv237. Epub 2015 Nov 2. PMID 26525063
- [Background] Fagerstrom KO. Can reduced smoking be a way for smokers not interested in quitting to actually quit? Respiration. 2005 Mar-Apr;72(2):216-20. doi: 10.1159/000084057. PMID 15824536
- [Background] Grace RC, Kivell BM, Laugesen M. Gender differences in satisfaction ratings for nicotine electronic cigarettes by first-time users. Addict Behav. 2015 Nov;50:140-3. doi: 10.1016/j.addbeh.2015.06.027. Epub 2015 Jun 12. PMID 26135334
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Hecht SS. Oral Cell DNA Adducts as Potential Biomarkers for Lung Cancer Susceptibility in Cigarette Smokers. Chem Res Toxicol. 2017 Jan 17;30(1):367-375. doi: 10.1021/acs.chemrestox.6b00372. Epub 2016 Dec 1. PMID 28092948
- [Background] Hughes JR. The hardening hypothesis: is the ability to quit decreasing due to increasing nicotine dependence? A review and commentary. Drug Alcohol Depend. 2011 Sep 1;117(2-3):111-7. doi: 10.1016/j.drugalcdep.2011.02.009. Epub 2011 Mar 15. PMID 21411244
- [Background] Hughes JR, Hatsukami D. Signs and symptoms of tobacco withdrawal. Arch Gen Psychiatry. 1986 Mar;43(3):289-94. doi: 10.1001/archpsyc.1986.01800030107013. PMID 3954551
- [Background] Irwin DE, Atwood CA Jr, Hays RD, Spritzer K, Liu H, Donohue JF, Leidy NK, Yount SE, DeWalt DA. Correlation of PROMIS scales and clinical measures among chronic obstructive pulmonary disease patients with and without exacerbations. Qual Life Res. 2015 Apr;24(4):999-1009. doi: 10.1007/s11136-014-0818-1. Epub 2014 Oct 12. PMID 25307510
- [Background] King BA, Patel R, Nguyen KH, Dube SR. Trends in awareness and use of electronic cigarettes among US adults, 2010-2013. Nicotine Tob Res. 2015 Feb;17(2):219-27. doi: 10.1093/ntr/ntu191. Epub 2014 Sep 19. PMID 25239961
- [Background] Le Houezec J. Role of nicotine pharmacokinetics in nicotine addiction and nicotine replacement therapy: a review. Int J Tuberc Lung Dis. 2003 Sep;7(9):811-9. PMID 12971663
- [Background] Morean ME, Krishnan-Sarin S, Sussman S, Foulds J, Fishbein H, Grana R, O'Malley SS. Psychometric Evaluation of the E-cigarette Dependence Scale. Nicotine Tob Res. 2019 Oct 26;21(11):1556-1564. doi: 10.1093/ntr/ntx271. PMID 29301008
- [Background] Patel D, Davis KC, Cox S, Bradfield B, King BA, Shafer P, Caraballo R, Bunnell R. Reasons for current E-cigarette use among U.S. adults. Prev Med. 2016 Dec;93:14-20. doi: 10.1016/j.ypmed.2016.09.011. Epub 2016 Sep 7. PMID 27612572
- [Background] Peng Y, Croce CM. The role of MicroRNAs in human cancer. Signal Transduct Target Ther. 2016 Jan 28;1:15004. doi: 10.1038/sigtrans.2015.4. eCollection 2016. PMID 29263891
- [Background] Popova L, Ling PM. Alternative tobacco product use and smoking cessation: a national study. Am J Public Health. 2013 May;103(5):923-30. doi: 10.2105/AJPH.2012.301070. Epub 2013 Mar 14. PMID 23488521
- [Background] Rose M, Bjorner JB, Gandek B, Bruce B, Fries JF, Ware JE Jr. The PROMIS Physical Function item bank was calibrated to a standardized metric and shown to improve measurement efficiency. J Clin Epidemiol. 2014 May;67(5):516-26. doi: 10.1016/j.jclinepi.2013.10.024. PMID 24698295
- [Background] Shadel WG, Edelen MO, Tucker JS, Stucky BD, Hansen M, Cai L. Development of the PROMIS nicotine dependence item banks. Nicotine Tob Res. 2014 Sep;16 Suppl 3(Suppl 3):S190-201. doi: 10.1093/ntr/ntu032. PMID 25118226
- [Background] Shahab L, Goniewicz ML, Blount BC, Brown J, McNeill A, Alwis KU, Feng J, Wang L, West R. Nicotine, Carcinogen, and Toxin Exposure in Long-Term E-Cigarette and Nicotine Replacement Therapy Users: A Cross-sectional Study. Ann Intern Med. 2017 Mar 21;166(6):390-400. doi: 10.7326/M16-1107. Epub 2017 Feb 7. PMID 28166548
- [Background] Sobell, L., & Sobell, M. (1995). Alcohol consumption measures. In J. Allen & M. Columbus (Eds.), Assessing alcohol problems: A guide for clinicians and researcher (pp. 55-73). Bethesda, MD: National Institute on Alcohol Abuse & Alcoholism.
- [Background] Sobell, L., & Sobell, M. (2003). Alcohol consumption measures. In J. P. A. a. V. B. & Wilson (Eds.), Assessing alcohol problems: A guide for clinicians and researchers. (pp. 75-99). Bethesda, MD: National Institute on Alcohol Abuse & Alcoholism.
- [Background] Zhang M, Li G, Wang Y, Wang Y, Zhao S, Haihong P, Zhao H, Wang Y. PD-L1 expression in lung cancer and its correlation with driver mutations: a meta-analysis. Sci Rep. 2017 Aug 31;7(1):10255. doi: 10.1038/s41598-017-10925-7. PMID 28860576
- [Derived] Fucito LM, Baldassarri SR, Wu R, Gueorguieva R, Morean ME, Herbst RS, Krishnan-Sarin S, O'Malley SS. Effects of oral nicotine pouches on cigarette smoking behaviour and tobacco harm exposure: a randomised pilot trial in adults. Tob Control. 2025 Jun 23:tc-2024-059094. doi: 10.1136/tc-2024-059094. Online ahead of print. PMID 40550628

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.20 (9.70) | 55.47 (13.40) | 56.83 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Customized: Black/African American | 3 | 8 | 11
  Race Customized: White/Caucasian | 12 | 6 | 18
  Race Customized: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Smoke within 30 minutes of waking [Count of Participants; unit: Participants] — This is binary count of yes/no responses to whether or not participants smoke their first cigarette within 30 minutes of waking in the morning.
  Participants
    Yes | 10 | 10 | 20
    No | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Cigarettes Smoked Per Day (Log-transformed)
Description: The investigators will compare whether smoking behavior varies by the 3mg and 6mg nicotine concentrations as measure by the standardized Timeline Followback Interview.
Time Frame: up to week 4
Measure: Mean (Standard Deviation); unit: number of cigarettes smoked
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration
Number analyzed (Participants) | 15 | 15
number of cigarettes smoked | 2.0 (0.1) | 1.8 (0.1)

2. Secondary Outcome: Number of Participants Who Switched From Cigarettes to the ZYN Pouches.
Description: To investigate whether switching behavior varies by the 3mg and 6mg nicotine concentrations
Time Frame: This will be evaluated at week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration
Number analyzed (Participants) | 15 | 15
Participants | 0 | 2

3. Secondary Outcome: Percentage of Smoke Free Days.
Description: The investigators will compare whether the smoke free days vary by the 3mg and 6mg nicotine concentrations
Time Frame: up to week 4
Measure: Mean (Standard Deviation); unit: percentage of smoke free days
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration
Number analyzed (Participants) | 15 | 15
percentage of smoke free days | 8.57 (22.42) | 11.22 (24.58)
Statistical Analysis 1: Comparison: 3mg Nicotine Concentration vs 6mg Nicotine Concentration; Test type: Superiority; p = 0.601, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Level of Biomarker (NNAL) Among Smokers
Description: Participants will provide repeated lab samples for biomarker assessments. Urine samples obtained will be compared at baseline and week 4 for differences by group and by time.
Time Frame: baseline and week 4
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration
Number analyzed (Participants) | 15 | 15
pg/mL
  Baseline | 17.26 (1.89) | 15.98 (1.89)
  Week 4 | 18.55 (1.94) | 16.04 (1.91)

5. Secondary Outcome: Subjective Effects of Oral Nicotine Pouches
Description: To evaluate the acceptability of switching, participants will also be asked how likely it is that they will continue to use ZYN oral nicotine patches for cigarette substitution compared to cigarettes on a question designed for this trial.
Time Frame: week 4
Population: This measure was not used in the study and therefore data were not collected.
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | 3mg Nicotine Concentration | 6mg Nicotine Concentration
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 13/15 | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3mg Nicotine Concentration (N=15) | 6mg Nicotine Concentration (N=15)
chest pain (Cardiac disorders) | 1 | 1
rapid heartbeat (Cardiac disorders) | 1 | 3
vision problems (Eye disorders) | 1 | 1
abdominal pain (Gastrointestinal disorders) | 4 | 1
appetite changes (Gastrointestinal disorders) | 3 | 4
diarrhea (Gastrointestinal disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 4 | 6
vomiting (Gastrointestinal disorders) | 1 | 1
fatigue (General disorders) | 3 | 6
fever (General disorders) | 1 | 1
other (General disorders) | 6 | 8
sore throat (Infections and infestations) | 5 | 2
weight loss (Investigations) | 1 | 1
dizziness (Nervous system disorders) | 0 | 2
fainting (Nervous system disorders) | 0 | 0
headache (Nervous system disorders) | 7 | 6
vivid dreams (Psychiatric disorders) | 2 | 3
difficulty sleeping (Psychiatric disorders) | 4 | 3
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 | 3
coughing (Respiratory, thoracic and mediastinal disorders) | 5 | 5
itching or rash (Skin and subcutaneous tissue disorders) | 1 | 0
sweating (Skin and subcutaneous tissue disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT04250727/Prot_SAP_000.pdf